CLINICAL TRIAL: NCT04054362
Title: A Phase II Pilot Trial Of Paclitaxel Protein Bound and Gemcitabine Based Chemotherapy and the Addition Of Paricalcitol Upon Attainment of Stable or Progressive Disease in Patients With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Paricalcitol Addition to Chemotherapy in Patients With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: PINBALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012255
Record Dates: First submitted 2019-04-23; First posted 2019-08-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Taxes; Cisplatin; Gemcitabine; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Cisplatin (Experimental): Paclitaxel Protein bound, Cisplatin, and Gemcitabine until stable or progressive disease, at which point Paricalcitol will be introduced.
  Interventions: Drug: Paclitaxel protein bound; Drug: Cisplatin; Drug: Gemcitabine; Drug: Paricalcitol
- Without Cisplatin (Experimental): Paclitaxel Protein bound and Gemcitabine until stable or progressive disease, at which point Paricalcitol will be introduced.
  Interventions: Drug: Paclitaxel protein bound; Drug: Gemcitabine; Drug: Paricalcitol

INTERVENTIONS:
Drug: Paclitaxel protein bound — paclitaxel protein bound and gemcitabine with or without cisplatin until stable or progressive disease at which point paricalcitol will be introduced
Drug: Cisplatin — paclitaxel protein bound and gemcitabine with or without cisplatin until stable or progressive disease at which point paricalcitol will be introduced
  Arms: With Cisplatin
Drug: Gemcitabine — paclitaxel protein bound and gemcitabine with or without cisplatin until stable or progressive disease at which point paricalcitol will be introduced
Drug: Paricalcitol — paclitaxel protein bound and gemcitabine with or without cisplatin until stable or progressive disease at which point paricalcitol will be introduced

SUMMARY:
This is a phase II pilot trial of Paclitaxel Protein Bound and Gemcitabine based chemotherapy and the addition of Paricalcitol upon attainment of stable or progressive disease in eligible patients with untreated metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth-highest cancer killer worldwide with an overall 5 year survival of about 8%. The only potentially curative procedure, surgical excision, is feasible in a minority of patients, but even in these patients the majority (~80%) die within 5 years. This study aims to see if adding paricalcitol (a vitamin D analogue) to chemotherapy can slow down tumour growth in patients with previously untreated metastatic pancreatic cancer.

Studies have shown vitamin D can change the pancreatic tumour microenvironment from an immunologically suppressive (tumour growth promoting) to an immunologically hostile one, slowing down tumour growth in this way.

Patients with pancreatic cancer that has spread to other organs and who have adequate hepatic and renal function are eligible. Participants will receive chemotherapy (paclitaxel and gemcitabine, with or without cisplatin). On development of stable disease or disease progression, paricalcitol will be added to the chemotherapy regimen and participants will continue on this treatment until their cancer stops responding to treatment. After that participants will be followed up 3 monthly for the collection of disease status and survival data.

Participants will be asked to donate tumour and blood samples to allow the research team to look at the effects on the tumour biology.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Ability to comply with the protocol.
3. Aged ≥ 18 years; male or female.
4. Histologically or cytologically confirmed metastatic (stage IV) pancreatic ductal adenocarcinoma.
5. Karnofsky performance status ≥70.
6. At least one lesion that can be measured accurately at baseline as ≥10mm in the longest diameter (except lymph nodes which must have a short axis ≥15mm) with CT/MRI and which is suitable for repeated measurements per RECIST v1.1
7. Adequate haematological and end-organ function, as per the local institutions reference ranges, within 21 days prior to day 1 of cycle 1 of treatment defined by the following:

   1. Haematology: ANC >1.5 x 109/L (>1500 cells / mm3); Platelet count > 100 x 109/L (>100,000 cells/mm3); haematocrit level >27% for females or >30% for males
   2. Coagulation: INR and aPTT ≤1.5 x ULN.
   3. Biochemistry: serum creatinine < 1.5mg/dl, bilirubin < 1.5 x ULN; AST / ALT ≤ 2.5 x ULN (or ≤ 5 x ULN in the presence of liver metastasis) calculated creatinine clearance ≥ 50ml/min (as measured by Cockcroft & Gault)
8. Life expectancy ≥ 12 weeks.
9. Women of childbearing potential must agree not to become pregnant (e.g. post-menopausal for at least 1 year, surgically sterile, or using effective contraception) for the duration of the study and for 1 month after last dose of study treatment. Women of child bearing potential must have a negative serum or urine pregnancy test within 14 days of Cycle 1 Day 1 (preferably as close to the study treatment day as possible). Both male and female patients of reproductive potential must agree to use effective contraception from 2 weeks before the start of study treatment and until 6 month (female participants) or 6 months (male participants) after completion of treatment (as per protocol section 6.10.5).
10. Tumour sites amenable to repeated biopsies.
11. Willingness to undergo paired tumour biopsies during the trial

Exclusion Criteria:

1. Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatments in the adjuvant setting with gemcitabine and/or 5-FU or gemcitabine administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present. In exceptional circumstances, if a patient has received paclitaxel protein bound and gemcitabine as first line chemotherapy for metastatic disease in exactly the same way as mandated in the current trial, they can be considered eligible to be enrolled directly to the add on paricalcitol component of the trial.
2. Palliative surgery and/or radiation treatment less than 4 weeks prior to initiation of study treatment.
3. Exposure to any investigational agent within 4 weeks prior to initiation of study treatment.
4. Evidence of central nervous system (CNS) metastasis (negative imaging study, if clinically indicated, within 28 days of Cycle 1 Day 1).
5. History of other malignancies (except cured basal or squamous cell carcinoma, superficial bladder cancer, prostate cancer in active surveillance, or carcinoma in situ of the cervix) unless documented free of cancer for ≥2 years.
6. Current, serious, clinically significant cardiac arrhythmias as determined by the investigator.
7. History of HIV infection.
8. Active, clinically significant serious infection requiring treatment with antibiotics, antivirals or anti-fungals (see Section 6.10).
9. History of symptomatic genitourinary stones (e.g. kidney stones) within 12months of Cycle 1 Day 1.
10. Pre-existing, clinically significant peripheral neuropathy ≥ G2
11. Hypersensitivity to the active study drug substance or to any of its excipients as listed in section 6 of the SmPC of each study drug.
12. Patients with a history of pneumonitis
13. Patients with a history of a hearing impairment
14. Patients who have received any live vaccines within 4 weeks prior to trial registration
15. Patient is on prohibited concurrent medication (see Section 6.10). In particular, vitamin D and calcium supplements must be stopped at the time of enrolment and for the duration of study treatment.
16. Any other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of study treatment, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
17. Female patients who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Clinical benefit | Time frame will be measured from date of Paricalcitol until the date of documented progression or date of death from any cause, whichever came first, expected maximum length of 7 months.
  To determine the clinical benefit of adding paricalcitol to the regimens of either paclitaxel protein bound plus gemcitabine or paclitaxel protein bound plus cisplatin plus gemcitabine for patients with stable or progressive metastatic PDA.

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, London, Greater, United Kingdom

IPD SHARING:
Plan to Share IPD: No